CLINICAL TRIAL: NCT06044532
Title: SKAMo-1: Characterization of the Upper Layers of Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eclypia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-A02578-35
Record Dates: First submitted 2023-08-07; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin characterization (Experimental)
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Experimental — At the first visit, effects of skin preparations (cleaning or sanding) on skin parameters and wearing a sham device will be evaluated. At the second visit the effect on skin parameters of a local heating and an OGTT will be evaluated.

SUMMARY:
Diabetes is a frequent disease characterized by chronic hyperglycemia, and its prevalence is increasing worldwide. Historically, patients with diabetes were required to monitor capillary blood glucose concentration up to several times a day through fingertip sampling.

Recently marketed devices now allow measurements of interstitial fluid blood glucose continuously, thus limiting pain associated with sampling. However, they are still invasive and have to be changed every 14 days.

Therefore, to optimize continuous glycemia monitoring while avoiding pain, discomfort, and the risk of infection, non-invasive methods are needed. Among the different strategies being developed, optical wearable sensors with specific signal processing are a promising option. The sensors detecting this optical signal will be included in a device. Yet, wearing a device may slightly modify several properties of the skin, such as its humidity and thermal regulation, and subsequently have an impact on the measured optical signal. Therefore, it is important to better understand how a device affects these characteristics to include these parameters in the future device algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years and ≤ 60 years
* Signed informed consent
* Person who is affiliated to a social security scheme or who is beneficiary of such a scheme

Exclusion Criteria:

* Body mass index (BMI) > 30 kg/m2
* Any acute or chronic disease with vascular impact
* Any cutaneous disease on sites implicated in the study (dorsum of the forearm)
* Allergy to one of the material used in the sham device and during the procedure of the study
* The persons mentioned in articles L1121-5 to L1121-8 of the public health code may not be included in this research
* Subject who would receive more than 4500 euros in compensation due to his or her participation in other research involving the human person in the 12 months preceding this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Change of skin hydration on the dorsum of the forearm after two and a half hours of wearing the sham device. | Visit 1,Day 0, before and after two and a half hours of wearing the sham device
  Hydration is measured with a capacitance method, expressed as arbitrary units (dielectric value)

SECONDARY OUTCOMES:
Change of skin elasticity after the wearing the sham device | Visit 1,Day 0, before and after two and a half hours of wearing the sham device
  elasticity (suction method) expressed as penetration depth in mm/time
Change of transepidermal water loss after the wearing the sham device | Visit 1,Day 0, before and after two and a half hours of wearing the sham device
  transepidermal water loss (the density gradient of the water evaporation) expressed as the evaporation rate in g/h/m2
Change of thickness of the stratum corneum after the wearing the sham device | Visit 1,Day 0, before and after two and a half hours of wearing the sham device
  thickness of the stratum corneum (LC-OCT method) expressed as mm
Change of skin temperature after the wearing the sham device | Visit 1,Day 0, before and after two and a half hours of wearing the sham device
  skin temperature (infrared thermography) expressed as Celsius,
Change of skin blood flux after the wearing the sham device | Visit 1,Day 0, before and after two and a half hours of wearing the sham device
  skin blood flux (LSCI) expressed as an arbitrary unit,
Change of skin hydration after skin cleaning | Visit 1, Day 0, in 30 minutes, measures taken before and after skin cleaning
  expressed as previously described
Change of skin elasticity after skin cleaning | Visit 1, Day 0, in 30 minutes, measures taken before and after skin cleaning
  expressed as previously described
Change of transepidermal water loss after skin cleaning | Visit 1, Day 0, in 30 minutes, measures taken before and after skin cleaning
  expressed as previously described
Change of thickness of the stratum corneum after skin cleaning | Visit 1, Day 0, in 30 minutes, measures taken before and after skin cleaning
  expressed as previously described
Change of skin temperature after skin cleaning | Visit 1, Day 0, in 30 minutes, measures taken before and after skin cleaning
  expressed as previously described
Change of skin blood flux after skin cleaning | Visit 1, Day 0, in 30 minutes, measures taken before and after skin cleaning
  expressed as previously described
Change of skin hydration after skin sanding | Visit 1, Day 0, in 30 minutes, measures taken before and after skin sanding
  expressed as previously described
Change of skin elasticity after skin sanding | Visit 1, Day 0, in 30 minutes, measures taken before and after skin sanding
  expressed as previously described
Change of transepidermal water loss after skin sanding | Visit 1, Day 0, in 30 minutes, measures taken before and after skin sanding
  expressed as previously described
Change of thickness of the stratum corneum after skin sanding | Visit 1, Day 0, in 30 minutes, measures taken before and after skin sanding
  expressed as previously described
Change of skin temperature after skin sanding | Visit 1, Day 0, in 30 minutes, measures taken before and after skin sanding
  expressed as previously described
Change of skin blood flux after skin sanding | Visit 1, Day 0, in 30 minutes, measures taken before and after skin sanding
  expressed as previously described
Change of skin hydration after local heating | Visit 2, Day 7 (+/-6 days), before and after local heating (40 minutes local thermal heating between 33 to 43°C with probes PF457)
  expressed as previously described
Change of skin elasticity after local heating | Visit 2, Day 7 (+/-6 days), before and after local heating (40 minutes local thermal heating between 33 to 43°C with probes PF457)
  expressed as previously described
Change of transepidermal water loss after local heating | Visit 2, Day 7 (+/-6 days) before and after local heating (40 minutes local thermal heating between 33 to 43°C with probes PF457)
  expressed as previously described
Change of thickness of the stratum corneum after local heating | Visit 2, Day 7 (+/-6 days) before and after local heating (40 minutes local thermal heating between 33 to 43°C with probes PF457)
  expressed as previously described
Change of skin temperature after local heating | Visit 2, Day 7 (+/-6 days) before and after local heating (40 minutes local thermal heating between 33 to 43°C with probes PF457)
  expressed as previously described
Change of skin blood flux after local heating | Visit 2, Day 7 (+/-6 days) before and after local heating (40 minutes local thermal heating between 33 to 43°C with probes PF457)
  expressed as previously described
Change of skin hydration induced by oral glycemia tolerance test | Visit 2, Day 7 (+/-6 days), before and during oral glycemia tolerance test (every 15 minutes for 2 hours)
  expressed as previously described
Change of skin elasticity induced by oral glycemia tolerance test | Visit 2, Day 7 (+/-6 days), before and during oral glycemia tolerance test (every 15 minutes for 2 hours)
  expressed as previously described
Change of transepidermal water loss induced by oral glycemia tolerance test | Visit 2, Day 7 (+/-6 days), before and during oral glycemia tolerance test (every 15 minutes for 2 hours)
  expressed as previously described
Change of thickness of the stratum corneum induced by oral glycemia tolerance test | Visit 2, Day 7 (+/-6 days), before and during oral glycemia tolerance test (every 15 minutes for 2 hours)
  expressed as previously described
Change of skin temperature induced by oral glycemia tolerance test | Visit 2, Day 7 (+/-6 days), before and during oral glycemia tolerance test (every 15 minutes for 2 hours)
  expressed as previously described
Change of skin blood flux induced by oral glycemia tolerance test | Visit 2, Day 7 (+/-6 days), before and during oral glycemia tolerance test (every 15 minutes for 2 hours)
  expressed as previously described

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France